CLINICAL TRIAL: NCT06172829
Title: Clinical Validation of Suntech Advantage MX With Suntech Neonate and Children Cuff Line Against Invasive Intra-arterial Reference According to the ANSI/AAMI/ISO 810602-2019 Protocol for Neonates, Infants, Children
Brief Title: Clinical Validation of Suntech Advantage MX With Suntech Neonate and Children Cuff Line
Status: Withdrawn | Type: Observational
Why Stopped: no enrollment
Sponsor: SunTech Medical (Network)
Collaborators: Children's Hospital Los Angeles (Other)
Responsible Party: Sponsor
Other Study IDs: Advantage MX Neonate-Infant
Record Dates: First submitted 2023-11-30; First posted 2023-12-15 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Pediatric Postmarket Surveillance: Yes

GROUPS / COHORTS (5):
- At least 3 subjects shall be <1,000g in weight
  Interventions: Device: Advantage MX Module
- At least 3 subjects shall be 1,000g to 2,000g in weight
  Interventions: Device: Advantage MX Module
- At least 3 subjects shall be >2,000g
  Interventions: Device: Advantage MX Module
- At least 3 subjects shall be >/= 29 days and < 1 year of age
  Interventions: Device: Advantage MX Module
- At least 3 subjects shall be >/= 1 year and <3 years of age
  Interventions: Device: Advantage MX Module

INTERVENTIONS:
Device: Advantage MX Module — no intervention will be provided.

SUMMARY:
Patients will be selected according to specific criteria. Upon selection, patients with an existing intra-arterial line will have their blood pressure monitored with the SunTech Advantage MX module in addition to the reference data collected from intra-arterial line. Data collected from the Advantage MX module will be compared to the reference data from the intra-arterial line.

ELIGIBILITY:
Inclusion Criteria:

* At least 3 subjects shall be < 1,000g in weight.
* At least 3 subjects shall be 1,000g to 2,000g in weight.
* At least 3 subjects shall be >2,000g
* At least 3 subjects shall be ≥ 29 days and < 1 year of age.
* At least 3 subjects shall be ≥ 1 year and < 3 years of age.

Exclusion Criteria:

* Subjects who study personnel determine invasive blood pressure measurements will be unreliable
* Patients found to have a-fib, irregular heart rhythm, dysrhythmias, bigeminy, trigeminy, and isolated premature ventricular beats (VPBs) during the enrollment process are to be ineligibile to participate in the study
* Patients who are prescribed anti-coagulation medication during the enrollment process or begin anti-coagulation medication after enrollment are ineligible to participate in the study.
* Exclusions can also occur post-data review based on exclusion criteria according to ANSI/AAMI/ISO 81060-2:2019

Ages: 1 Month to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Study is only accepting neonate and pediatric patients who meet the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-11-07 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
The blood pressure measurement | approximately 1 hour
  collected from the Advantage MX module matches the intra-arterial line data

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided